CLINICAL TRIAL: NCT00455676
Title: Chevron Osteotomy Versus SCARF Osteotomy in the Treatment of Hallux Valgus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Limoges (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: I06020
Record Dates: First submitted 2007-04-03; First posted 2007-04-04 (Estimated); Last update posted 2008-12-30 (Estimated); Status verified 2008-12

CONDITIONS: Hallux Valgus
Keywords: Scarf Osteotomy; Chevron Osteotomy; Comparison
MeSH Terms: conditions — Hallux Valgus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Chevron osteotomy versus Scarf osteotomy

SUMMARY:
Comparison between two techniques of osteotomy wich are more or less invasive : two criterias : clinical data and x-rays data.

All patients operated for hallux valgus for 01/01/99 to 31/12/03 in the department of bone surgery CHU Limoges :

* Scarf or Jonhson (chevron) osteotomy
* Experienced surgeon : Pr ARNAUD, Pr MABIT or Pr CHARISSOUX.

DETAILED DESCRIPTION:
Prospective assessmentfor all patients with an average follow up of 5 years :

* Groulier score scale (similar to AOFAS score rating)
* X-rays data
* Clinical evaluation
* Pedoscopic data.

ELIGIBILITY:
Inclusion Criteria:

* All patients operated for hallux valgus for 01/01/99 to 31/12/03 in the department of bone surgery CHU Limoges.

  * Scarf or Johnson (Chevron) osteotomy,
  * Experienced surgeon : Pr MABIT, Pr ARNAUD, Pr CHARISSOUX.
* Age of Patients > 18 years.

Exclusion Criteria:

* Hallux valgus wich wasn't operated by these surgeons.
* No consentment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74
Dates: Start 2006-06; Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Comparison between two techniques of osteotomy wich are more or less invasive : two criterias : clinical data and x-rays data.

SECONDARY OUTCOMES:
Extension of chevron osteotomy indication. Check of results for one-year more operated patients by chevron osteotomy.
Comparaison of both techniques concerning post-operative complication.
Search of significative difference about satisfaction of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Chistrian MABIT, MD, Principal Investigator — CHU Limoges
Locations (1):
- Department of Bone Surgery, Limoges, France